CLINICAL TRIAL: NCT00583557
Title: A Multi-Center, Open-Label, Continuation Trial of LymphoStat-B™ Antibody (Monoclonal Anti-BLyS Antibody) in Subjects With Rheumatoid Arthritis (RA) Who Completed the Phase 2 Protocol LBRA01
Brief Title: A Continuation Trial for Subjects With Rheumatoid Arthritis That Have Completed Protocol LBRA01
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision - not related to safety
Sponsor: Human Genome Sciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LBRA99
Record Dates: First submitted 2007-12-20; First posted 2007-12-31 (Estimated); Results first posted 2011-06-29 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; RA
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — belimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Belimumab (Experimental)
  Interventions: Drug: belimumab

INTERVENTIONS:
Drug: belimumab — IV 10mg/kg Q28 days
  Other Names: LymphoStat-B™

SUMMARY:
This is a continuation trial of LymphoStat-B™ to evaluate the long-term safety in subjects with Rheumatoid Arthritis that completed study LBRA01 and benefitted from treatment.

DETAILED DESCRIPTION:
This is a multi-center, open label, continuation trial of LymphoStat-B™ in Rheumatoid Arthritis (RA) subjects who achieved at least an ACR20 response in the Phase 2 study LBRA01 (NCT00071812).

ELIGIBILITY:
Primary Inclusion Criteria:

1. Have completed the LBRA01 trial.
2. Have achieved at least an ACR20 response at the end of LBRA01.

Primary Exclusion Criteria:

1. Have switched NSAIDs due to worsening RA disease activity, used more than 10 mg/day of oral prednisone, or were given a corticosteroid injection during the last 30 days of LBRA01.
2. Required a new DMARD (not otherwise excluded in protocol LBRA01) to replace an ineffective one, or an additional DMARD (not to exceed 2 DMARDs in total) within the last 60 days of LBRA01.
3. Used prohibited medications during their participation in LBRA01. These medications include the following:

   * Other investigational agents.
   * Biologic response modifiers
   * Cyclophosphamide.
   * Corticosteroid injections (except 1 injection of up to 40 mg of prednisone into an inflamed joint or intramuscularly every 6 months).
   * 2 new DMARDs.
   * 1 new DMARD plus high dose prednisone >10 mg/day.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2005-01; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (48):
- United States (44):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - Arizona Arthritis Research, Paradise Valley, Arizona
  - Arthritis Health, Scottsdale, Arizona
  - The University of Arizona Health Sciences Center, Tucson, Arizona
  - University of Southern CA, Los Angeles, California
  - Wallace Rheumatic Disease Center, Los Angeles, California
  - Boling Clinical Trials, Rancho Cucamonga, California
  - Arthritis Care Center, Inc., San Jose, California
  - Arthritis Associates & Osteoporosis Center of Colorado Springs, Colorado Springs, Colorado
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Arthritis and Rheumatic Disease Specialties, Aventura, Florida
  - Rheumatology Associates of Central Florida, Orlando, Florida
  - Tampa Medical Group, P.A., Tampa, Florida
  - Radiant Research Boise, Boise, Idaho
  - Rheumatology Associates, Chicago, Illinois
  - Medical Specialists, Munster, Indiana
  - Kentuckiana Center for Better Bone and Joint Health, Louisville, Kentucky
  - The Osteoporosis and Arthritis Clinical Trial Center, Cumberland, Maryland
  - Center for Rheumatology and Bone Research, Wheaton, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Washington University in St. Louis, St Louis, Missouri
  - Arthritis Center of Nebraska, Lincoln, Nebraska
  - Strafford Medical Associates, P.A., Dover, New Hampshire
  - The Center for Rheumatology, Albany, New York
  - North Shore University Hospital, Manhasset, New York
  - Arthritis Clinic and Carolina Bone and Joint, Charlotte, North Carolina
  - Wake Forest Unviersity School of Medicine, Winston-Salem, North Carolina
  - Bone and Joint Hospital - Research Department, Oklahoma City, Oklahoma
  - Oklahoma Medical Reseach Foundation, Oklahoma City, Oklahoma
  - Oklahoma Center for Arthritis Therapy & Research, Tulsa, Oklahoma
  - University of Pittsburgh School of Medicine & ASPH, Pittsburgh, Pennsylvania
  - Rheumatic Disease Associates, Willow Grove, Pennsylvania
  - Arthritis Centers of Texas, Dallas, Texas
  - UT Southwestern Medical Center at Dallas, Dallas, Texas
  - Houston Institute for Clinical Research, Houston, Texas
  - Texas Research Center, Sugar Land, Texas
  - IPC Clinical Research, Ogden, Utah
  - Arthritis Clinic of Northern Virginia, P.C., Arlington, Virginia
  - Seattle Arthritis Clinic, Seattle, Washington
  - Arthritis Northwest Rheumatology, Spokane, Washington
  - Rheumatology Northwest Clinical Trials, Yakima, Washington
  - Rheumatic Disease Center, Glendale, Wisconsin
  - Gundersen Clinic, LTD, La Crosse, Wisconsin
  - Marshfield Medical Research Foundation, Wausau, Wisconsin
- Poland (4):
  - NZOZ Centrum Medyczne, Bialystok
  - Wojewodzki Zespol Reumatologiczny, Sopot
  - Instytut Reumaologii, Warsaw
  - Instytut Reumatologii, Warsaw

REFERENCES:
- See also: ClinicalTrials.gov Posting for Parent Protocol LBRA01 — http://clinicaltrials.gov/ct2/show/NCT00071812?term=lbra01&rank=2

RESULTS

PARTICIPANT FLOW:
Groups:
- Belimumab 10 mg/kg: Subjects received belimumab at a dose of 10 mg/kg IV every 28 days for up to 5 years in this protocol
Period: Overall Study
Arm/Group | Belimumab 10 mg/kg
Started | 155
Received at Least 1 Dose Belimumab | 153
Completed | 85 (Completer defined as subjects whose reason for discontinuation was sponsor discontinuation of study)
Not Completed | 70
Not completed — Withdrawal by Subject | 18
Not completed — Adverse Event | 9
Not completed — Lack of Efficacy | 31
Not completed — Lack of Compliance | 5
Not completed — Other | 5
Not completed — Did not receive belimumab in LBRA99 | 2

BASELINE CHARACTERISTICS:
Arm/Group | Belimumab 10 mg/kg
Number analyzed (Participants) | 153
Age Continuous [Mean (Standard Deviation); unit: years] | 51.1 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118
  Male | 35

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate the Long-term Safety of LymphoStat-B™ in Subjects With RA.
Description: SEE ALSO ADVERSE EVENT (AE) RESULTS SECTION.
Time Frame: Up to 5 years
Measure: Number; unit: Particpants
Arm/Group | Belimumab 10 mg/kg
Number analyzed (Participants) | 153
Particpants
  Number of subjects with at least 1 AE | 148
  Number of subjects with at least 1 Non-Serious AE | 144
  Number of subjects with at least 1 Serious AE | 47
  Number of subjects with an AE resulting in death | 3

2. Secondary Outcome: The Efficacy Endpoints Will Include Long-term ACR Responses, DAS28 Response, C-reactive Protein (CRP), Erythrocyte Sedimentation Rate (ESR), and Rheumatoid Factor (RF).
Description: NOT ANALYZED
Time Frame: up to 5 Years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 5 years
Description: Subjects in LBRA99 completed parent study LBRA01 (NCT00071812) during which they received belimumab (1, 4 or 10 mg/kg belimumab) for 6 mos or 1 yr.
Arm/Group | Belimumab 10 mg/kg
Serious Adverse Events (participants affected / at risk) | 47/153
Other Adverse Events (participants affected / at risk) | 144/153
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Belimumab 10 mg/kg (N=153)
Anaemia (Blood and lymphatic system disorders) | 3
Angina pectoris (Cardiac disorders) | 3
Arteriosclerosis coronary artery (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 2
Coronary artery thrombosis (Cardiac disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Colitis ulcerative (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Diverticulum intestinal (Gastrointestinal disorders) | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Hiatus hernia (Gastrointestinal disorders) | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Obstruction gastric (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Non-cardiac chest pain (General disorders) | 2
Cholecystitis acute (Hepatobiliary disorders) | 1
Appendicitis perforated (Infections and infestations) | 1
Bacterial pyelonephritis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Epiglottitis (Infections and infestations) | 1
Escherichia bacteraemia (Infections and infestations) | 1
Gastritis bacterial (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 2
Gastroenteritis viral (Infections and infestations) | 1
Incision site infection (Infections and infestations) | 1
Laryngitis fungal (Infections and infestations) | 1
Meningitis pneumococcal (Infections and infestations) | 1
Mycobacterium avium complex infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 3
Pyelonephritis (Infections and infestations) | 2
Sepsis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Dislocation of vertebra (Injury, poisoning and procedural complications) | 1
Head injury (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Weight decreased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Hand deformity (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2
Joint instability (Musculoskeletal and connective tissue disorders) | 2
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 6
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebellar infarction (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Cervicobrachial syndrome (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Lumbar radiculopathy (Nervous system disorders) | 1
Movement disorder (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 2
Major depression (Psychiatric disorders) | 1
Obsessive-compulsive disorder (Psychiatric disorders) | 1
Acute prerenal failure (Renal and urinary disorders) | 1
Cervical dysplasia (Reproductive system and breast disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Accelerated hypertension (Vascular disorders) | 1
Peripheral ischaemia (Vascular disorders) | 1
Vascular insufficiency (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Belimumab 10 mg/kg (N=153)
Anaemia (Blood and lymphatic system disorders) | 10
Abdominal pain (Gastrointestinal disorders) | 9
Diarrhoea (Gastrointestinal disorders) | 24
Dyspepsia (Gastrointestinal disorders) | 13
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 12
Nausea (Gastrointestinal disorders) | 16
Vomiting (Gastrointestinal disorders) | 14
Fatigue (General disorders) | 21
Oedema peripheral (General disorders) | 28
Seasonal allergy (Immune system disorders) | 16
Bronchitis (Infections and infestations) | 35
Gastroenteritis viral (Infections and infestations) | 11
Influenza (Infections and infestations) | 15
Nasopharyngitis (Infections and infestations) | 18
Sinusitis (Infections and infestations) | 39
Tooth abscess (Infections and infestations) | 9
Upper respiratory tract infection (Infections and infestations) | 53
Urinary tract infection (Infections and infestations) | 23
Viral upper respiratory tract infection (Infections and infestations) | 21
Contusion (Injury, poisoning and procedural complications) | 8
Excoriation (Injury, poisoning and procedural complications) | 9
Skin laceration (Injury, poisoning and procedural complications) | 12
Weight increased (Investigations) | 10
Hypercholesterolaemia (Metabolism and nutrition disorders) | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 66
Back pain (Musculoskeletal and connective tissue disorders) | 31
Bursitis (Musculoskeletal and connective tissue disorders) | 8
Joint swelling (Musculoskeletal and connective tissue disorders) | 24
Muscle spasms (Musculoskeletal and connective tissue disorders) | 11
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 20
Myalgia (Musculoskeletal and connective tissue disorders) | 11
Neck pain (Musculoskeletal and connective tissue disorders) | 10
Osteopenia (Musculoskeletal and connective tissue disorders) | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 36
Rheumatoid nodule (Musculoskeletal and connective tissue disorders) | 10
Synovitis (Musculoskeletal and connective tissue disorders) | 11
Dizziness (Nervous system disorders) | 13
Headache (Nervous system disorders) | 23
Depression (Psychiatric disorders) | 15
Insomnia (Psychiatric disorders) | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 27
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 8
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 9
Rash (Skin and subcutaneous tissue disorders) | 9
Tooth extraction (Surgical and medical procedures) | 14
Hypertension (Vascular disorders) | 23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For multi-center trials, no investigator will be authorized to publish study results from an individual center until the earlier of the multi-center trial results are published or 12 months after the end or termination of the multi-center trial at all sites. All manuscripts and abstracts must be submitted to the sponsor for review least 30 days prior to submission for publication or for presentation at a scientific meeting. The sponsor may delay publication for up to 3 months.